CLINICAL TRIAL: NCT06753825
Title: Comparison of the Efficacy of Transcutaneous Pulsed Radiofrequency Therapy and Calcium Channel Blockers in Childhood Migraine Headache.
Brief Title: Childhood Migraine Treatment Noninvasive Pulsed Radiofrequency vs Flunarizine
Status: Active, not recruiting | Type: Observational
Sponsor: Damla Yürük (Other)
Responsible Party: Sponsor-Investigator, Damla Yürük, medical doctor, Diskapi Teaching and Research Hospital
Organization: Diskapi Teaching and Research Hospital (Other)
Other Study IDs: childhood migraine treatment
Record Dates: First submitted 2024-12-30; First posted 2024-12-31 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Migraine Disease
MeSH Terms: interventions — Flunarizine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group pulsed radiofrequency: The group receiving pulsed radiofrequency therapy via transcutaneous electrodes receives 2 sessions of treatment, each lasting 8 minutes, once a week.
  Interventions: Device: Radiofrequency
- group medical teratment: The group receiving 5 mg flunarizine treatment per day
  Interventions: Drug: flunarizine

INTERVENTIONS:
Device: Radiofrequency — radiofrequency treatment
  Groups: group pulsed radiofrequency
Drug: flunarizine — flunarizine oral treatment
  Groups: group medical teratment

SUMMARY:
The aim of this observational study was to investigate the long-term effects of patients receiving interventional transcutaneous electrode-pulsed radiofrequency therapy versus calcium channel blockers for the treatment of childhood migraine pain. The main question to be answered was.

Which of the long-term effects of interventional transcutaneous pulsed radiofrequency versus calcium channel blockers for the treatment of childhood migraine pain is more effective? Participants who have started both treatments will answer questions about their headaches in an online survey for 3 months as part of their regular medical care.

DETAILED DESCRIPTION:
There are two groups in the trial. One group will receive transcutaneous pulsed radiofrequency treatment for a total of 3 weekly sessions. The other group will receive 1x 5 mg flunarizine active ingredient. Both groups will consist of 30 patients. All patients will be followed from the start of treatment and will be assessed at month 1 and month 3 using the paediatric migraine disability index, headache diaries and visual pain scale.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with migraine according to ICHD-3 Migraine criteria
* Being between the ages of 8-18
* Having 4 or more migraine attacks per month

Exclusion Criteria:

* Other primary or secondary headache diagnosis
* Patient could not be reached during follow-up

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Total 60 patients, per group 30 patients
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Headache diary | month 1 and month 3
  The headache diary : including the date, triggering event, severity (rated on a scale from 1-very mild- to 5-very severe-), type, location of the pain. Additional symptoms such as nausea, vomiting, light sensitivity, sound sensitivity, and dizziness and duration of the pain, and whether daily activities were impacted are recorded.

SECONDARY OUTCOMES:
Pediatrik migraine disability scale PedMidas | month 1 and month 3
  PedMIDAS is a validated questionnaire consisting of six questions designed to assess the impact of headaches on the daily functioning of children and adolescents over the past three months. The form evaluates the extent to which headaches have affected school attendance, academic performance, ability to complete homework, and participation in family, social, and recreational activities. Respondents are asked to report the number of days missed or days when they functioned at less than half of their normal capability in these areas. A high score was associated with increased disability. If the PedMIDAS score was between 0-10, the disability was considered 'not - very mild', between 11-30 was considered 'mild', between 31-50 was considered 'moderate', 51 and above was considered 'severe'

CONTACTS AND LOCATIONS:
Locations (1):
- Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No